CLINICAL TRIAL: NCT00153023
Title: A Prospective, Randomised, Double-blind, Double-dummy, Forced-titration, Multicentre, Parallel Group, One Year Treatment Trial to Investigate the Efficacy of Telmisartan 80 mg Versus Valsartan 160 mg in Hypertensive Type 2 Diabetic Patients With Overt Nephropathy VIVALDI-Study
Brief Title: 1 Year Trial Telmisartan 80 mg Versus Valsartan 160 mg in Hypertensive Type 2 Diabetic Patients With Overt Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.396
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Diabetic Nephropathies; Hypertension
MeSH Terms: conditions — Diabetic Nephropathies; Hypertension | interventions — Telmisartan; Valsartan

INTERVENTIONS:
Drug: Telmisartan
Drug: Valsartan

SUMMARY:
The general aim of this study is to compare telmisartan 80 mg with valsartan 160 mg in hypertensive patients with type 2 diabetes and overt nephropathy with adjusted blood pressure beyond the target of 130/80 mmHg after one year of treatment.

The primary objective of this study is to show that telmisartan 80 mg is at least as effective (i.e., not inferior) and possibly superior to valsartan 160 mg in reducing 24 hour proteinuria after one year of treatment.

DETAILED DESCRIPTION:
This is a randomised, double-blind, double-dummy, forced titration, multicentre, parallel group trial in patients with essential hypertension, diabetes mellitus type 2 and diabetic nephropathy.

After a 4-6 week Run-in period, patients are randomised to one of the treatment groups and receive either Telmisartan 40 - 80 mg or Valsartan 80 - 160 mg. The treatment regimen is a forced titration with the lower dose given for 2 weeks and the higher dose given for the rest of the treatment period summing up to 52 weeks of treatment. During the treatment period, 8 visits to the investigator are scheduled in order to control blood pressure, renal function parameters and safety. In addition, parameters of endothelial function and oxidative stress are measured at baseline, 6 months and after one year of treatment.

Study Hypothesis:

Non-inferiority of telmisartan 80 mg compared to valsartan 160 mg will be tested using the following set of hypotheses:

Null Hypothesis:

The overall mean change from baseline in UPER (24 hour urinary protein excretion rate) for telmisartan 80 mg is inferior to that for valsartan 160 mg by 0.5 g/day or more.

Alternative Hypothesis:

The overall mean change from baseline in UPER (24 hour urinary protein excretion rate) for telmisartan 80 mg is less than 0.5 g/day worse than that for valsartan 160 mg.

Comparison(s):

In order to test the non-inferiority hypothesis, analysis of covariance with treatment and centre as main effects and baseline as a covariate will be performed. Time-to-event data will be analysed using the log-rank test.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus
2. Aged 30-70 years of age
3. Hypertension at screening defined as:

   * an average cuff systolic blood pressure > 130 mmHg and/or diastolic blood pressure >80 mmHg in untreated patients OR
   * patients receiving antihypertensive therapy (i.e., medications specifically prescribed to treat hypertension)
4. Overt nephropathy defined by 24 hour proteinuria >= 900 mg and by serum creatinine below 265 mol/l (3.0 mg/dl)

Exclusion Criteria: None

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885
Dates: Start 2003-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12

PRIMARY OUTCOMES:
Change from baseline (Visit 6) in 24 hour proteinuria, after one year of treatment (study end) with telmisartan 80 mg versus valsartan 160 mg. | Baseline, after 1 year of treatment

SECONDARY OUTCOMES:
Change from baseline in 24-hour urinary albumin excretion rate (UAER). | Baseline, after 1 year of treatment
Change from baseline in 24-hour urinary sodium excretion rate. | Baseline, after 1 year of treatment
Change from baseline in serum creatinine. | Baseline, after 1 year of treatment
Change from baseline in creatinine clearance | Baseline, after 1 year of treatment
Change from baseline in estimated glomerular filtration rate (eGFR). | Baseline, after 1 year of treatment
Change from baseline in plasma asymmetrical dimethylarginine (ADMA) levels. | Baseline, after 1 year of treatment
Change from baseline in urine 8-iso-prostaglandin F2α levels | Baseline, after 1 year of treatment
Change from baseline in serum high sensitive C-reactive protein (CRP) levels. | Baseline, after 1 year of treatment
Time to a composite of a doubling of serum creatinine concentration , end-stage renal disease (ESRD), or all cause death | after 1 year of treatment
Time to a composite of morbidity and mortality from cardiovascular causes (myocardial infarction (MI), stroke, first hospitalisation for heart failure or unstable angina, coronary or peripheral revascularisation). | after 1 year of treatment
Change from baseline in insulin sensitivity (Homeostasis Model Assessment (HOMA) index). | Baseline, after 1 year of treatment
Change from baseline in plasma adiponectin levels. | Baseline, after 1 year of treatment
Change from baseline in BP endpoints (SBP, DBP and pulse pressure) | Baseline, after 1 year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (109):
- Czechia (7):
  - University Hospital St. Anna, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Vihohrady, Prague
  - General University Hospital, Prague
  - District Hospital Tabor, Tábor
  - Masaryk Hospital, Ústí nad Labem
  - Hospital Usti nad Orlici, Ústí nad Orlicí
- Denmark (5):
  - Medical Department, Copenhagen NV
  - Medicinsk afdeling, Fredericia
  - Medicinsk afdeling F, Endokrinologisk, Hiller?d
  - Endokrinologisk afdeling, Hvidovre
  - Medical Department, Roskilde
- France (11):
  - Chu Sud, Amiens
  - Centre Hospitalier, Beauvais
  - Hopital Duchenne, Boulogne-sur-Mer
  - Hopital Clemenceau, Caen
  - Centre Hospitalier, Dunkirk
  - Hopital Albert Michalon, La Tronche
  - Hopital A.Mignot, Le Chesnay
  - Hopital Maison Blanche, Reims
  - Hopital Yves Le Foll, Saint-Brieuc
  - Hopital Saint Quentin, Saint-Quentin
  - Centre Hospitalier, Valenciennes
- Germany (18):
  - Boehringer Ingelheim Investigational Site, Aschaffenburg
  - Diabetes Klinik Bad Mergentheim, Bad Mergentheim
  - Institut fur Klinische Forschung, Berlin
  - Charite Campus Buch, Berlin
  - KFH Dialysezentrum, Eberswalde
  - Universitatsklinik Heidelberg, Heidelberg
  - Boehringer Ingelheim Investigational Site, Karlsruhe
  - Institut fur Klinische Forschung, Mainz
  - Boehringer Ingelheim Investigational Site, Münster
  - Boehringer Ingelheim Investigational Site, Neuwied
  - Boehringer Ingelheim Investigational Site, Pirna
  - Boehringer Ingelheim Investigational Site, Riesa
  - Boehringer Ingelheim Investigational Site, Rosenheim
  - Boehringer Ingelheim Investigational Site, Saarbrücken
  - Boehringer Ingelheim Investigational Site, Saarlouis
  - Boehringer Ingelheim Investigational Site, Sinsheim
  - Boehringer Ingelheim Investigational Site, Speyer
  - Internist, Würzburg
- Italy (10):
  - Azienda Ospedaliera Policlinico S. Orsola Malpighi, Bologna
  - Ospedali Riuniti di Livorno, Livorno
  - Presidio Ospedaliero Campo di Marte, Lucca
  - Universita degli Studi "Federico II", Napoli
  - Azienda Ospedaliera di Padova, Padua
  - IRCCS Policlinico S.Matteo, Pavia
  - Policlinico Monteluce, Perugia
  - Azienda Ospedaliera S. Maria degli Angeli, Pordenone
  - Ospedale "S. Maria delle Croci", Ravenna
  - Universita Tor Vergata, Roma
- Malaysia (6):
  - Penang General Hospital, George Town
  - Hospital Ipoh, Ipoh, Perak
  - University Sains Malaysia, Kelantan
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Putrajaya, Kuala Selangor
- Portugal (9):
  - Centro Hospitalar de Coimbra, Coimbra
  - Hospital Distrital de Faro, Faro
  - Hospital Curry Cabral, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Hospital de Santa Marta, Lisbon
  - Associac?o Protectora dos Diabeticos de Portugal, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital de S. Jo?o, Porto
  - Centro Hospitalar Vila Nova de Gaia, Vila Nova de Gaia
- Russia (10):
  - Medical Academy named Sechenova I.M., Moscow
  - Russian State Medical University, Moscow
  - National Endocrinology Research Center of Russia, Moscow
  - President's Medical Center, Moscow
  - Russian Cardiology Research Center, Moscow
  - Russian Academy for Advanced Medical Studies, Moscow
  - Moscow President's Medical Center, Moscow
  - Regional Clinical Scientific Research Institute, Moscow
  - City Hospital of Saint Elizaveta, Saint Petersburg
  - Military Medical Academy, Saint Petersburg
- Slovakia (10):
  - NovaMed, Banská Bystrica
  - Ministry Hospital of Internal Affairs, Bratislava
  - Faculty Hospital, Bratislava
  - Faculty Hospital of L. Derer, Bratislava
  - Diabetologic and Internal Clinic, Lučenec
  - Faculty Hospital, Nitra
  - Hospital Nove Mesto, Nové Mesto
  - Regional Hospital Nove Zamky, Nové Zámky
  - MSP-DIAGNOSTIK, Ltd., Trenčín
  - Faculty Hospital Trnava, Trnava
- South Korea (2):
  - Keimyung University Dongsan Medical Center, Daegu
  - Yonsei University Medical Center, Seoul
- Spain (9):
  - Hospital Torrecardenas, Almería
  - Hospital Ntra. Sra de Sonsoles, Ávila
  - Hospital Clinico y Provincial de Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital de Cabuenes, Gijón
  - Hospital Virgen del Rocio, Seville
  - Hospital Universitario La Fe, Valencia
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Chi Mei Medical Center, Dawan
  - Buddhist Tzu Chi Hospital, Hualien City
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
- Ukraine (7):
  - Dnyepropyetrovsk Medical Academy, Dnyepropetrovsk
  - Kharkiv Medical State University, Kharkiv
  - Institute of Diabetic pathology problems, Kharkiv
  - Institute of Cardiology, Kiev
  - V.P. Komisarenko Institute of Endocrinology and Metabolism, Kiev
  - Kyiv Clinical Hospital No. 1, Kyiv
  - Zaporozhye Regional Clinical Hospital, Zaporizhzhya